CLINICAL TRIAL: NCT04595435
Title: Prospective Registry of Intraoperative Radiation Therapy Using Low Energy X-ray for Breast Cancer at Medical Center, Navicent Health
Brief Title: IORT-Breast at Medical Center Navicent Health
Acronym: IORT-Breast
Status: Active, not recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Navicent (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00092014; H1901940 (Other: Medical Center Central Georgia IRB); IORT (Other: Atrium Health Navicent)
Record Dates: First submitted 2019-04-08; First posted 2020-10-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Female; Early-stage Breast Cancer
Keywords: Intraoperative Radiation Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Cohort A- Preoperative Prospective: Subjects are eligible to receive IORT and have agreed to participate in the study prior to any intervention.
  Interventions: Procedure: Lumpectomy; Radiation: Intraoperative Radiation Therapy
- Cohort B- Postoperative Prospective: Subjects who have had IORT performed within the previous 6 month who agree to participate.
  Interventions: Procedure: Lumpectomy; Radiation: Intraoperative Radiation Therapy

INTERVENTIONS:
Procedure: Lumpectomy — Removal of lump/tumor from breast utilizing an approach that saves as much breast as possible.
  Other Names: Breast Conserving Surgery
Radiation: Intraoperative Radiation Therapy — Delivery of low energy radiation therapy directly at surgical site, immediately removal of lump and tissue prior to final surgical closure
  Other Names: IORT

SUMMARY:
Intraoperative Breast Radiation Therapy (IORT-Breast) utilizing the Xoft Axxent Electronic Brachytherapy System (Xoft) has been recently introduced as a treatment option for women 50 years of age and older who have early stage, low risk Invasive Breast Cancer (IBC). Clinical trials have shown IORT to be non-inferior to whole breast radiation, however some concern continues with rates of recurrence and clinical outcomes.

Given the recent introduction and continued debate it is an excellent opportunity to observe and monitor outcomes in the patients that are treated at Navicent Health through this prospective, observational registry. The opportunity also permits examination of the participant's thoughts and feeling on Quality of Life and Cosmetic Appearance

DETAILED DESCRIPTION:
Objectives: (primary and important secondary objectives) The primary objective is to determine rates of recurrence at 5, and 10 years following IORT-Breast at Navicent Health.

Secondary objectives include determination of acute and late effects of IORT-Breast at the treatment site, cosmetic outcomes and satisfaction over 10 years.

In addition, the study will determine why patients who were scheduled for IORT-Breast did not receive it after lumpectomy.

Study Design:

Prospective, observational registry.

Setting/Participants:

The study focuses on outpatients/short stay surgery performed at the Medical Center, Navicent Health, Macon, GA only.

Participants have been deemed eligible for IORT-Breast or have received IORT-Breast within the last 6 months. Key eligibility criteria for IORT- Breast includes women, aged 55 years old or greater, diagnosed with clinically node negative, grade 1 or 2 Invasive Breast Cancer with no lymphovascular invasion, that is 20mm or less in greatest dimension, Estrogen Receptor (ER) positive, HER 2 Neu Negative, and with a depth greater than 10mm from skin.

Study Interventions and Measures:

Participants will be eligible for IORT-Breast or have received IORT-Breast in the previous 6 months. Participants who were scheduled for IORT-Breast and do not receive IORT-Breast will have reasons for not receiving IORT-Breast recorded and will not be followed further. Participants receiving IORT-Breast will have treatment parameters recorded and will be followed every 6 months for 2 years and then annually until up to 10 years following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and HIPAA authorization
* T1 tumor (less than or equal to 20mm in greatest diameter)
* Unifocal
* Histological Grade 1 or 2
* Node Negative
* ER +ve
* HER-2 -ve

Exclusion Criteria:

* Previous radiation therapy to the involved breast other than IORT within 6 months
* High grade tumors (Histologic grade 3)
* Her-2 Positive
* Lymphovascular invasion
* Metastatic disease
* close proximity to or involvement of skin
* Multifocal cancer

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at Navicent Health who meet eligibility criteria for IORT-Breast or who have received IORT-Breast within the previous 6 months
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrence | 5 year
  To determine rate of recurrence of disease at specific time period
Rate of recurrence | 10 year
  To determine rate of recurrence of disease at specific time period

SECONDARY OUTCOMES:
Acute and late effects | 5 years
  To determine the rate of acute and late effects of IORT at the treatment site. Periodic review by surgeon and self reports identifying acute and late effects and calculating the rate of incidence for the treated group.
Treatment Abandonment | 5 years
  To determine rate and reason for abandoning procedure after being scheduled for procedure. Calculating the rate of those who were scheduled to receive IORT and then did not receive the treatment as planned and reason why they did not receive the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dale, MD, Principal Investigator — Atrium Health Navicent Physician's Group; David Cole, MD, Principal Investigator — Central Georgia Radiation Oncology
Locations (1):
- Medical Center, Navicent Health, Macon, Georgia, United States

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT04595435/Prot_ICF_000.pdf